CLINICAL TRIAL: NCT05980845
Title: The Effect of Nature Sounds and Music on Vital Signs and Anxiety Levels of Hemodialysis Patients
Brief Title: The Effect Nature Sounds and Music on Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, IMarasli, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12.09.2018-4
Record Dates: First submitted 2023-07-10; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Hemodialysis Complication; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Interventions (Active Comparator): It was explained to the patients in the nature sounds group that nature sounds would be played for 30 minutes in three HD sessions for one week, starting from the beginning of the session. Afterwards, the patients were informed about the usage of the Mp3 player and in-ear headphones, they were demonstrated that they could adjust the volume to the level they desired, and it was stated that they should not detach the headphones until the 30-minute recording was over. The patients listened to nature sounds for 30 minutes in three HD sessions for one week under the supervision of the researcher.
  Interventions: Behavioral: Nature sounds
- Control Group (No Intervention): Patients in the control group were not intervened by the researcher during the HD sessions. Before the first HD session started, the "Descriptive Characteristics Form" and "Trait Anxiety Scale" were performed by the researcher while the patients were in the waiting room. Then, in every three HD sessions for one week, when the patients went to their beds, their vital signs were measured and recorded on the "Vital Signs Monitoring Form" and the "State Anxiety Scale" was administered just before the HD treatment session was started. Then, the vital signs of the patients were measured and recorded on the "Vital Signs Monitoring Form" at the 30th minute, 1st, 2nd, 3rd hour of the HD session and immediately after the end of the HD session. At the same time, the "State Anxiety Scale" was performed again immediately after the end of the HD session. The patient was then transferred out of the unit.

INTERVENTIONS:
Behavioral: Nature sounds — Nature sounds would be played for 30 minutes in three HD sessions for one week, starting from the beginning of the session. Afterwards, the patients were informed about the usage of the Mp3 player and in-ear headphones, they were demonstrated that they could adjust the volume to the level they desired, and it was stated that they should not detach the headphones until the 30-minute recording was over.
  Other Names: music
  Arms: Assigned Interventions

SUMMARY:
The study was conducted as a randomized controlled experimental research to examine the effect of nature sounds and music on vital signs and anxiety levels of hemodialysis patients.

The study was conducted between September 6, 2019 and March 21, 2020 with 75 patients who received treatment in the hemodialysis units of three hospitals, one university, one education research and one state hospital in Antalya province, met the inclusion criteria and consented to participate in the study. Patients were homogenously divided into intervention (nature sound group n=25 and music group n=25) and control (n=25) groups on the basis of age, gender and hemodialysis duration. Patients in the intervention group were subjected to nature sounds/music during the hemodialysis procedure, while patients in the control group were not subjected to any intervention during the procedure. The data were collected by face-to-face interview technique using the "Descriptive Characteristics Form", "Vital Signs Monitoring Form", "State Anxiety Inventory" and "Trait Anxiety Inventory". Ethics committee approval, institutional permissions and written consent of the patients were obtained for the implementation of the study. Number, percentage, mean, standard deviation, minimum and maximum, the the Shapiro Wilk normality test, One-Way Analysis of Variance, Chi-Square tests, the Kruskal Wallis test, Dunn-Bonferroni test, Tukey HSD, Three-Way Analysis of Variance and Bonferroni Corrected Two Ratio Z test were employed in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Age range between 18 and 79,
* Receiving HD treatment for at least six months,
* Receiving three sessions of HD treatment per week on a regular outpatient basis at the same institution.

Exclusion Criteria:

* Any problem that prevents cognitive, affective and verbal communication,
* Having any psychiatric condition,
* Use of anxiolytic medication,
* Out of the criteria for inclusion in the study,

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale (SAS) | Change in anxiety score during Nature Sounds and Music, an average of 10 minutes
  State Anxiety Scale (SAS) is used to determine how an individual feels at a certain moment and under certain conditions. According to the degree of severity of the emotions, thoughts or behaviors expressed by the items, "not at all" (1), "a little" (2), "a lot" (3), "completely" (4) in the scale. Some of the items in the scale are direct statements and some of them are reversed statements.
The Trait Anxiety Scale (TAS) | Change in anxiety score during Nature Sounds and Music, an average of 10 minutes
  The Trait Anxiety Scale (TAS) is used to determine how the individual usually perceives themselves. The items are scored as "almost never" (1), "sometimes" (2), "very often" (3) and "almost always" (4) according to the frequency of the feelings, thoughts or behaviors expressed by the items. The items in the scale are in the form of direct and inverted statements.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Hagemann PMS, Martin LC, Neme CMB. The effect of music therapy on hemodialysis patients' quality of life and depression symptoms. J Bras Nefrol. 2019 Jan-Mar;41(1):74-82. doi: 10.1590/2175-8239-jbn-2018-0023. Epub 2018 Sep 13. PMID 30222176
- [Result] Kim Y, Evangelista LS, Park YG. Anxiolytic Effects of Music Interventions in Patients Receiving Incenter Hemodialysis: A Systematic Review and Meta-Analysis. Nephrol Nurs J. 2015 Jul-Aug;42(4):339-47; quiz 348. PMID 26462307